CLINICAL TRIAL: NCT01197950
Title: A Randomized Controlled Trial of Acupuncture to Reduce Labour Pain
Brief Title: Acupuncture With Manual and Electrical Stimulation to Reduce Labour Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Skövde (Other)
Responsible Party: Principal Investigator, Lena B Martensson, PhD RNM Senior Lecturer, University of Skövde
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 136-08
Record Dates: First submitted 2010-08-26; First posted 2010-09-09 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Labour Pain
Keywords: acupuncture; labour; pain; pain relief; complementary
MeSH Terms: conditions — Labor Pain; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual Acupuncture (Active Comparator): Manual stimulation
  Interventions: Device: Manual Acupuncture
- Electro Acupuncture (Experimental): Electrical and manual stimulation
  Interventions: Device: Electro Acupuncture
- Standard care (No Intervention): No acupunture

INTERVENTIONS:
Device: Manual Acupuncture — The women will receive treatment on bilateral points, both distal points and local points and the needles will be manually stimulated to reach De Qi every ten minutes during one hour.
  Other Names: Acupuncture
  Arms: Manual Acupuncture
Device: Electro Acupuncture — The women will receive treatment on bilateral points, both distal points and local points and the needles will be manually stimulated to reach De Qi every ten minutes during one hour. Eight needles in the painful area (local points) will be connected to an electro-stimulator and stimulated with high frequency (80 Hz) square wave pulses (0.18-ms duration) with alternating polarity. The woman will adjust the intensity of the electrical stimulation to be just under pain threshold.
  Other Names: Acupuncture
  Arms: Electro Acupuncture

SUMMARY:
The purpose of this study is to evaluate the effect of manual acupuncture and electro-acupuncture on labour pain.

DETAILED DESCRIPTION:
Acupuncture is used in obstetric care in spite of insufficient evidence of its potential to reduce labour pain. The findings so far are contradictory, which may reflect methodological limitations. The present study will take issues into account, such as sufficiently large sample to allow detection of possible differences between study groups; optimal timing of the intervention; controlling for intensity of the treatment; qualified training of persons giving the treatment; biological markers of pain and stress; possible effects on mother and infant; women's experiences such as overall birth experience and memory of pain.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the labour ward in spontaneous onset of labour
* Latent or active phase of labour
* Nulliparity
* Singleton pregnancy, cephalic presentation
* Gestation: 37+0 to 41+6 (weeks + days)
* Expressed need for labour pain relief
* Swedish speaking (well enough to understand written and oral instructions)

Exclusion Criteria:

* No pharmacological pain relief within 24 hours prior to inclusion into the study
* Severe preeclampsia
* Treatment with oxytocin at the time point of allocation
* Treatment with anticoagulant
* Pacemaker

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena B Martensson, PhD, Principal Investigator — University of Skövde
Locations (1):
- School of Life Sciences, University of Skövde, Skövde, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vixner L, Martensson LB, Schytt E. Acupuncture with manual and electrical stimulation for labour pain: a two month follow up of recollection of pain and birth experience. BMC Complement Altern Med. 2015 Jun 12;15:180. doi: 10.1186/s12906-015-0708-2. PMID 26066641
- [Background] Vixner L, Martensson LB, Stener-Victorin E, Schytt E. Manual and electroacupuncture for labour pain: study design of a longitudinal randomized controlled trial. Evid Based Complement Alternat Med. 2012;2012:943198. doi: 10.1155/2012/943198. Epub 2012 Apr 17. PMID 22577468
- [Background] Vixner L, Schytt E, Martensson LB. Associations between maternal characteristics and women's responses to acupuncture during labour: a secondary analysis from a randomised controlled trial. Acupunct Med. 2017 Jun;35(3):180-188. doi: 10.1136/acupmed-2016-011164. Epub 2016 Dec 16. PMID 27986648
- [Background] Vixner L, Schytt E, Stener-Victorin E, Waldenstrom U, Pettersson H, Martensson LB. Acupuncture with manual and electrical stimulation for labour pain: a longitudinal randomised controlled trial. BMC Complement Altern Med. 2014 Jun 9;14:187. doi: 10.1186/1472-6882-14-187. PMID 24913704

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Standard Care No acupucture
Period: Overall Study
Arm/Group | Manual Acupuncture | Electro Acupuncture | Standard Care
Started | 99 | 103 | 101
Completed | 83 (women's request (9), high workload (3), returned home (1), partus in one hour (1), other (2)) | 87 (women's request (11) high workload (4) returned to home (1)) | 83 (woman's request (11) high workload (1) returned to home (2) other (4))
Not Completed | 16 | 16 | 18
Not completed — Women's request (31), high workload (8), returned home (4), partus in one hour (1), other (6) | 16 | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Acupuncture | Electro Acupuncture | Standard Care | Total
Number analyzed (Participants) | 99 | 103 | 101 | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 99 | 103 | 101 | 303
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 103 | 101 | 303
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 99 | 103 | 101 | 303

OUTCOME MEASURES:

1. Primary Outcome: Use of Epidural Analgesia
Description: Frequecy of epidural analgesia
Time Frame: From start of treatment until birth
Measure: Number; unit: participants
Groups:
- Standard Care: Standard care
Arm/Group | Manual Acupuncture | Electro Acupuncture | Standard Care
Number analyzed (Participants) | 99 | 103 | 101
participants | 99 | 103 | 101

ADVERSE EVENTS:
Time Frame: Three hours
Description: We did not expected any adverse event except for infections in the injection area or after the acupuncture needles were removed.
Groups:
- Standard Care: Standard care - no acupuncture treatment at all
Arm/Group | Manual Acupuncture | Electro Acupuncture | Standard Care
All-Cause Mortality (participants affected / at risk) | 99/99 | 103/103 | 101/101
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/103 | 0/101
Other Adverse Events (participants affected / at risk) | 0/99 | 0/103 | 0/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Acupuncture (N=99) | Electro Acupuncture (N=103) | Standard Care (N=101)
Only minor adverse events were expected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No